CLINICAL TRIAL: NCT00869752
Title: A Phase I-II Trial of MK-0646, a Monoclonal Antibody Against Insulin-Like Growth Factor-1 Receptor, in Combination With Etoposide and Cisplatin in Extensive Stage Small Cell Lung Cancer
Brief Title: MK-0646, Etoposide, and Cisplatin in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I190; CAN-NCIC-IND190 (Registry Identifier: NCI US - Physician Data Query); CDR0000634447 (Other: PDQ)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: combined type small cell lung cancer; fusiform type small cell lung cancer; polygonal type small cell lung cancer; lymphocyte-like type small cell lung cancer; extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — dalotuzumab; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): MK-0646, a monoclonial antibody in combination with etoposide and cisplatin.
  Interventions: Biological: anti-IGF-1R recombinant monoclonal antibody MK-0646; Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Biological: anti-IGF-1R recombinant monoclonal antibody MK-0646 — MK-0646 should be given 1st followed within 30-60 minutes by cisplatin and then etoposide for cycles which include both MK-0646 and chemotherapy. Cycles are 21 days
Drug: cisplatin — MK-0646 should be given 1st followed within 30-60 minutes by cisplatin and then etoposide for cycles which include both MK-0646 and chemotherapy. Cycles are 21 days
Drug: etoposide — MK-0646 should be given 1st followed within 30-60 minutes by cisplatin and then etoposide for cycles which include both MK-0646 and chemotherapy. Cycles are 21 days

SUMMARY:
RATIONALE: Monoclonal antibodies, such as MK-0646, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as etoposide and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I/II trial is studying the side effects and best dose of MK-0646 when given together with etoposide and cisplatin and to see how well it works in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the recommended phase II dose of MK-0646 in combination with a standard etoposide and cisplatin chemotherapy regimen in patients with extensive stage small cell lung cancer. (phase I)
* To assess the toxicity and tolerability of this regimen in these patients. (phases I and II)
* To evaluate the preliminary efficacy of this regimen in these patients. (phase I)
* To assess the efficacy of this regimen, in terms of objective response rate, as well as complete response rate in these patients. (phase II)
* To assess progression-free survival and overall survival of patients treated with this regimen. (phase II)
* To explore the predictive and prognostic impact of biomarkers in patients treated with this regimen. (phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of MK-0646 followed by a phase II study.

Patients receive MK-0646 IV over 1 hour on days 1, 8, and 15 and cisplatin IV and etoposide IV once daily on days 1-3. Treatment repeats every 3 weeks for 4 to 8 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients with complete response (CR) or partial response (PR) may continue MK-0646 in the absence of disease progression, with temporary discontinuation while undergoing prophylactic cranial irradiation or thoracic radiotherapy.

Blood samples are collected at baseline (pre-dose) and periodically for biomarker and pharmacogenetic correlative studies. Blood samples are analyzed for changes in expression of IGF biomarkers (e.g., IGF-1, IGF-2 and IGF-PB), haplotype tagging analysis of the IGF-1R, and evaluation of the immunoglobulin G fragment C receptor polymorphisms.

After completion of study therapy, patients are followed at 4 weeks. Patients with responding disease (i.e., CR, PR, or stable disease) are followed every 3 months until relapse or progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)

  * Extensive stage disease that is incurable but amenable to treatment with platinum-based chemotherapy
  * Small cell and variant histologies allowed
  * No mixed tumors (i.e., small and large cell) or other neuroendocrine tumors of the lung
* Clinically and/or radiologically documented measurable disease, defined as ≥ 1 unidimensionally measurable site of disease ≥ 20 mm by chest x-ray, ≥ 15 mm by CT scan (lymph nodes), or ≥ 10 mm by CT scan or physical exam
* No uncontrolled or symptomatic CNS metastases

  * Patients who have completed radiotherapy or have undergone complete resection of CNS metastases are allowed provided they are on stable (non-increasing) or decreasing doses of corticosteroids

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 12 weeks
* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN (≤ 5 times ULN if documented liver metastases)
* Serum creatinine ≤ ULN OR creatinine clearance ≥ 50 mL/min
* Not pregnant or lactating
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after completion of study therapy
* No other active cancer
* No untreated and/or uncontrolled cardiovascular or other comorbid conditions

  * Patients with a significant cardiac history, even if controlled, should have a LVEF > 50%
* No uncontrolled diabetes
* Must be accessible for treatment and follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior cytotoxic chemotherapy or other IGF-1R targeting agents for SCLC
* At least 3 weeks since prior radiotherapy to neurological sites
* No prior radiotherapy to the lungs
* Prior surgery allowed provided that wound healing has occurred

  * At least 14 days since prior major surgery
* No other concurrent investigational agents or therapy
* No other concurrent anticancer treatment
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12-16 (Actual); Primary Completion 2012-03-15 (Actual); Study Completion 2012-07-04 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of MK-0646 in combination with standard etoposide and cisplatin chemotherapy | Each dose level
  Evaluate safety, tolerability in combination with standard chemotherapy.
Toxicity and tolerability according to NCI CTCAE v3.0 | Phase 1, each dose level and Phase II
  Look at toxicity and tolerability of MK0646 in combination with standard therapy.
Preliminary efficacy | Phase 1 dose levels, evey other cycle
  Look for evidence of response
Objective response rate | Phase II portion, every other cycle
  Determine objective response rate including complete response rate, progression free survival and overall survival.
Predictive and prognostic impact of biomarkers | Each cycle
  Blood samples will be collected and analyzed for occurrence of human-anti-humanized antibody response to MK0646 as well as IGF-1R analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ellis, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (3):
- Canada (3):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] J Clin Oncol 30, 2012 (suppl; abstr 7093)
- [Result] Ellis PM, Shepherd FA, Laurie SA, Goss GD, Olivo M, Powers J, Seymour L, Bradbury PA. NCIC CTG IND.190 phase I trial of dalotuzumab (MK-0646) in combination with cisplatin and etoposide in extensive-stage small-cell lung cancer. J Thorac Oncol. 2014 Mar;9(3):410-3. doi: 10.1097/JTO.0000000000000058. PMID 24518092